CLINICAL TRIAL: NCT06821646
Title: Social Cognition in Major Depression and Autism Spectrum Disorder: Cortical Excitatory-inhibitory Imbalance and Neuromechanism
Brief Title: Investigating the Brain's Physiological Responses in Depression and Autism, Using Transcranial Magnetic Stimulation and Electroencephalography
Status: Enrolling by invitation | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Other Study IDs: 202209019DINB
Record Dates: First submitted 2025-02-03; First posted 2025-02-12 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-12

CONDITIONS: Autism; Major Depressive Disorder (MDD)
Keywords: Autism; Major Depressive Disorder; FEPPA PET; TMS-EEG
MeSH Terms: conditions — Autistic Disorder; Depressive Disorder, Major | interventions — Positron-Emission Tomography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Autism
  Interventions: Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: transcranial magnetic stimulation and electroencephalography(TMS-EEG)
- Major Depression Disorder
  Interventions: Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: transcranial magnetic stimulation and electroencephalography(TMS-EEG)
- Autism, Major Depression Disorder
  Interventions: Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: transcranial magnetic stimulation and electroencephalography(TMS-EEG)
- Typically Developing Control
  Interventions: Diagnostic Test: Positron Emission Tomography (PET); Diagnostic Test: transcranial magnetic stimulation and electroencephalography(TMS-EEG)

INTERVENTIONS:
Diagnostic Test: Positron Emission Tomography (PET) — 18F-N-((2-(2-(fluoro-18f)ethoxy)phenyl)methyl)-N-(4-phenoxy-3-pyridinyl) acetamide
Diagnostic Test: transcranial magnetic stimulation and electroencephalography(TMS-EEG) — single pulse and paired pulse

SUMMARY:
The goal of this observational study is to investigate the brain physiological responses in depression and autism. The main questions aim to answer are:

1. Comparing the ratios of cortical excitation and inhibition among four groups: autism group, autism with depression group, depression group, and normal control group using Transcranial magnetic stimulation and electroencephalography (TMS-EEG). This study explores the relationship between the ratios of cortical excitation and inhibition and the severity of clinical symptoms.
2. Comparing the brain inflammation among four groups: autism group, autism with depression group, depression group, and normal control group using Positron emission tomography (PET). This study investigates the relationship between brain inflammation and the severity of clinical symptoms.
3. The mutual influence between the severity of brain inflammation and Excitatory/inhibitory imbalance (E/I imbalance).

Participants will receive clinical assessment, neurocognitive function tests, TMS-EEG, gamma oscillation, and PET examinations.

ELIGIBILITY:
Inclusion Criteria:

* Autism group : Adults aged 20-50 diagnosed with autism spectrum disorder。Intelligence Quotient(IQ) > 70, with autonomous abilities.
* Autism group with comorbid depression : Adults aged 20-50 diagnosed with autism spectrum disorder. Diagnosed with depression. IQ > 70. Not on antidepressants for at least one week, with autonomous abilities.
* Major depression disorder group : Adults aged 20-50. Diagnosed with major depressive disorder according to Diagnostic and Statistical Manual of Mental Disorders-IV-TR(DSM-IV-TR). IQ > 70. Not on antidepressants for at least one week, with autonomous abilities.
* Typically developing control group : Adults aged 20-50. Never diagnosed with autism spectrum disorder. Never diagnosed with depression. IQ > 70, with autonomous abilities.

Exclusion Criteria:

* Previously diagnosed with bipolar disorder, schizophrenia, attention deficit hyperactivity disorder (ADHD), or substance use disorder according to DSM-IV.
* Previously suffered from major medical or neurological diseases.
* Brain structural abnormalities (e.g., brain tumor or arteriovenous malformations) or neurological diseases (e.g., meningitis, encephalitis, stroke, or epilepsy).
* Previously undergone or soon to undergo brain surgery, or have metal implants in the head or neck area, such as neuro-stimulators or cochlear implants.
* Have a cardiac pacemaker.
* Pregnant participants.
* Participants with strong suicidal intentions.
* Other conditions that render the patient unable to cooperate, such as unsuitability after screening, unstable physical illness, or refusal to sign the informed consent.
* Claustrophobia, unable to undergo positron emission tomography(PET) and functional magnetic resonance imaging (fMRI) scans.
* Taking medications that may affect Excitatory/inhibitory balance (E/I balance).

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 160 (Estimated)
Dates: Start 2024-05-28 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Standardized Uptake Value (SUV) of Translocator Protein activity imaged by Positron Emission Tomography (PET) | 1 hour
Standardized Uptake Value (SUV) of Translocator Protein activity recorded by transcranial magnetic stimulation and electroencephalography(TMS-EEG) | 2 hours

SECONDARY OUTCOMES:
the total composite scores of multiple scales | 2 hours
  Adult Autism Spectrum Quotient (AQ), Empathy Quotient(EQ), Social Responsiveness Scale(SRS), Beck Depression Inventory(BDI), Beck Anxiety Inventory(BAI), The Schutte's Emotion Intelligence Scale(SEIS), Depression and Somatic Symptoms Scale(DSSS), Snaith-Hamilton Pleasure Scale(SHAPS)

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided